CLINICAL TRIAL: NCT00439374
Title: A Randomized Trial of 17 Alpha-Hydroxyprogesterone Caproate for Prevention of Preterm Birth in Nulliparous Women With a Short Cervix
Brief Title: RCT of Progesterone to Prevent Preterm Birth in Nulliparous Women With a Short Cervix
Acronym: SCAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Halted by NICHD after recommendation by DSMC to stop for futility
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HD36801 SCAN; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD053097 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD034136 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD036801 (NIH); U10HD053118 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Preterm Delivery; Cervical Length
Keywords: nulliparous; pregnancy; short cervix; progesterone
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Intervention Model Description: Treatment with 17 alpha-hydroxyprogesterone caproate via weekly injections of 250 mg of 17p until 37 weeks gestation or delivery vs. weekly injections of placebo oil until 37 weeks gestation or delivery.
Who Masked: Participant, Care Provider
Masking Description: Patients and care providers are masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 17 alpha-hydroxyprogesterone caproate (Active Comparator): 250 mg of 17 alpha-hydroxyprogesterone caproate given by weekly injection until 37 weeks gestation or delivery
  Interventions: Drug: 17 alpha-hydroxyprogesterone caproate
- Placebo (Placebo Comparator): Placebo oil given by weekly injection until 37 weeks gestation or delivery.
  Interventions: Other: Placebo Oil

INTERVENTIONS:
Drug: 17 alpha-hydroxyprogesterone caproate — Coded study medication is sterile solution containing 250 mg/mL of 17 alpha-hydroxyprogesterone caproate in castor oil with benzyl benzoate and benzyl alcohol as a preservative; placebo is same without the active ingredient. Study drug is administered as weekly 1 ml intramuscular injections until 36 week 6 days of gestation or delivery, whichever occurs first.
  Other Names: 17 AHP
  Arms: 17 alpha-hydroxyprogesterone caproate
Other: Placebo Oil — Placebo oil is a 250 mg/mL solution of castor oil with benzyl benzoate and benzyl alcohol as a preservative
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if giving progesterone medication to pregnant women, who have never delivered a baby after 19 weeks of pregnancy and who have a short cervix, lowers the risk of early delivery and improves the health of their baby.

DETAILED DESCRIPTION:
Preterm births, defined as the delivery of a baby less than 37 weeks of gestation, are responsible for the majority of neonatal mortality and morbidities. Studies have shown that a number of risk factors, including never having a baby before and having a short cervix are associated with early delivery. Recently the NICHD did a study in women who were pregnant again after having delivered preterm. It showed that giving 17 alpha-hydroxyprogesterone caproate (17P) medication during pregnancy decreased the chance of delivering another preterm baby by 34%. This placebo-controlled randomized clinical trial will address the primary research question: does treatment with 17P initiated before 23 weeks of gestation prevent delivery prior to 37 weeks in nulliparous women with a singleton gestation who have a short cervix?

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Cervical length as measured on transvaginal examination < 30mm between gestational ages of 16 weeks 0 days to 22 weeks 3 days
* Gestational age 16 weeks 3 days to 22 weeks 6 days at time of randomization

Exclusion Criteria:

* Multifetal gestation
* Progesterone treatment after 14 weeks 6 days during current pregnancy
* Vaginal bleeding, heavier than spotting, after 15 weeks 6 days
* Amniotic membranes prolapsed beyond external os
* Preterm rupture of membranes
* Fetal anomaly
* Pregnancy without a viable fetus
* Current or planned cervical cerclage
* Congenital Mullerian abnormality of the uterus
* Contraindication to intra-muscular injections
* Hypertension requiring medication
* Diabetes managed with insulin or oral hypoglycemic agents
* DES exposure
* Cervical surgery such as cold knife conization
* Planned indicated preterm delivery
* Participation in another interventional study that influences age at delivery
* Participation in this trial in a previous pregnancy
* Prenatal care or delivery planned outside a MFMU Network center

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Grobman, MD, MBA, Principal Investigator — Northwestern University; Menachem Miodovnik, MD, Study Director — NICHD Project Scientist
Locations (14):
- United States (14):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University-Prentice Hospital, Chicago, Illinois
  - Dept of OB/GYN, Hutzel Hospital, Detroit, Michigan
  - Columbia University-St. Luke's Hospital, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve-Metrohealth, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - University of Pittsburgh-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University -Women and Infants Hospital, Providence, Rhode Island
  - Dept of OB/GYN, Southwestern Medical Center, University of Texas, Dallas, Texas
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - University of Texas-Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses. Requests for datasets can be sent to mfmudatasets@bsc.gwu.edu

REFERENCES:
- [Derived] Grobman WA, Thom EA, Spong CY, Iams JD, Saade GR, Mercer BM, Tita AT, Rouse DJ, Sorokin Y, Wapner RJ, Leveno KJ, Blackwell S, Esplin MS, Tolosa JE, Thorp JM Jr, Caritis SN, Van Dorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. 17 alpha-hydroxyprogesterone caproate to prevent prematurity in nulliparas with cervical length less than 30 mm. Am J Obstet Gynecol. 2012 Nov;207(5):390.e1-8. doi: 10.1016/j.ajog.2012.09.013. Epub 2012 Sep 17. PMID 23010094
- See also: Click here for more information about the SCAN protocol — http://www.bsc.gwu.edu/mfmu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2007 through May 2011, the fourteen centers of the Maternal-Fetal Medicine Units Network of the Eunice Kennedy Shriver National Institute of Child Health and Human Development participated in this randomized double-blind placebo-controlled trial. Eligible women were offered participation.
Pre-assignment Details: Women who signed informed consent received a "compliance" injection of the placebo and were asked to return at least 3 days later for randomization. If a woman did not return for a randomization visit before 23 weeks 0 days of gestation, she was excluded.
Groups:
- 17 Alpha-hydroxyprogesterone Caproate: 17 alpha-hydroxyprogesterone caproate
  17 alpha-hydroxyprogesterone caproate : Coded study medication is sterile solution containing 250 mg/mL of 17 alpha-hydroxyprogesterone caproate in castor oil with benzyl benzoate and benzyl alcohol as a preservative; placebo is same without the active ingredient. Study drug is administered as weekly 1 ml intramuscular injections until 36 week 6 days of gestation or delivery, whichever occurs first.
- Placebo: castor oil
Period: Overall Study
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Started | 327 | 330
Completed | 327 | 330
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo | Total
Number analyzed (Participants) | 327 | 330 | 657
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (5.3) | 21.6 (4.4) | 22.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 330 | 657
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 76 | 74 | 150
  Non-hispanic black | 179 | 161 | 340
  Hispanic white | 19 | 38 | 57
  Hispanic black | 2 | 0 | 2
  Asian | 4 | 3 | 7
  Other | 47 | 54 | 101
Prepregnancy body mass index [Mean (Standard Deviation); unit: kg^m2] | 26.1 (6.9) | 25.4 (6.5) | 25.7 (6.7)
Prior Pregnancy [Count of Participants; unit: Participants]
  <13 wk of gestation | 92 | 82 | 174
  13-19 wk of gestation | 13 | 10 | 23
Payment for obstetric care [Count of Participants; unit: Participants]
  Uninsured/self-pay | 17 | 30 | 47
  Private insurance | 74 | 62 | 136
  Government-assisted insurance | 236 | 238 | 474
Married or living with partner [Count of Participants; unit: Participants] | 125 | 110 | 235
Alcohol use during pregnancy [Count of Participants; unit: Participants] | 33 | 20 | 53
Smoking during pregnancy [Count of Participants; unit: Participants] | 48 | 62 | 110
Illicit substance use during pregnancy [Count of Participants; unit: Participants] | 15 | 24 | 39
Gestational age at randomization [Mean (Standard Deviation); unit: weeks] | 21.4 (1.2) | 21.3 (1.3) | 21.4 (1.3)
Cervical length at screening [Mean (Standard Deviation); unit: mm] | 23.9 (5.6) | 23.8 (5.7) | 23.8 (5.7)
Cervical length at screening <15mm [Count of Participants; unit: Participants] | 25 | 31 | 56
Cervical funnel present [Count of Participants; unit: Participants] | 88 | 69 | 157
Cervical funnel length [Mean (Standard Deviation); unit: mm] — Population: Includes only the patients that had a cervical funnel present.
  mm
    number analyzed (Participants) | 88 | 69 | 157
    (all) | 14.8 (8.0) | 16.7 (8.7) | 15.6 (8.4)
Debris present [Count of Participants; unit: Participants] | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Delivering Before 37 Weeks Gestation
Description: Number of participants delivering before 37 weeks gestation by indication
Time Frame: Delivery before 37 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants
  Total Delivery <37 wk | 82 | 80
  Spontaneous | 54 | 55
  Medically indicated | 27 | 25
  Fetal loss/abortion <20 wk | 1 | 0
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; All deliveries less than 37 weeks; Test type: Superiority or Other; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.79 to 1.35]
Statistical Analysis 2: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Spontaneous deliveries; Test type: Superiority or Other; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.70 to 1.40]
Statistical Analysis 3: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Medically-indicated deliveries; Test type: Superiority or Other; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.65 to 1.84]

2. Secondary Outcome: Mean Gestational Age at Delivery
Description: Mean gestational age at delivery
Time Frame: Delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
weeks | 37.6 (3.9) | 37.4 (4.3)
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants With Preterm Premature Rupture of Membranes
Time Frame: <37 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants | 25 | 24
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.61 to 1.80]

4. Secondary Outcome: Number of Participants Who Delivered Before 35 Weeks Gestation
Description: Delivery before 35 weeks gestation
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants | 44 | 53
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.58 to 1.21]

5. Secondary Outcome: Number of Participants Who Delivered Before 32 Weeks Gestation
Description: Delivery before 32 weeks gestation
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants | 28 | 32
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.54 to 1.43]

6. Secondary Outcome: Number of Participants Who Delivered Before 28 Weeks Gestation
Description: Delivery before 28 weeks gestation
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants | 15 | 22
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.69, 95% CI 2-sided [0.36 to 1.30]

7. Secondary Outcome: Number of Participants Who Visited the Hospital Due to Preterm Labor
Description: Number of participants who visited the hospital due to preterm labor before 37 weeks gestation
Time Frame: Between randomization and 37 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants | 145 | 151
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.82 to 1.15]

8. Secondary Outcome: Number of Participants Who Underwent Tocolytic Therapy
Description: Number of participants who underwent tocolytic therapy during pregnancy
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 6 participants in the treatment group and 5 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 321 | 325
Participants | 35 | 42
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.55 to 1.29]

9. Secondary Outcome: Number of Participants Who Underwent Corticosteroid Therapy
Description: Number of participants who underwent corticosteroid therapy in pregnancy
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 6 participants in the treatment group and 5 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 321 | 325
Participants | 55 | 51
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.77 to 1.55]

10. Secondary Outcome: Number of Participants Who Had a Cerclage Placement
Description: Number of participants who had a cerclage placement
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 6 participants in the treatment group and 5 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 321 | 325
Participants | 6 | 4
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.52, 95% CI 2-sided [0.43 to 5.33]

11. Secondary Outcome: Number of Participants Experiencing Gestational Hypertension or Preeclampsia
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 1 participant in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 329
Participants | 46 | 40
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.78 to 1.72]

12. Secondary Outcome: Number of Participants With Gestational Diabetes Mellitus
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants | 15 | 13
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.56 to 2.41]

13. Secondary Outcome: Number of Participants Experiencing Cholestasis
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 1 participant in the Placebo group
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 329
Participants | 1 | 0

14. Secondary Outcome: Number of Participants Who Experienced Placental Abruption
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 328
Participants | 11 | 15
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.34 to 1.58]

15. Secondary Outcome: Number of Participants Who Experienced Chorioamnionitis
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 328
Participants | 29 | 20
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.45, 95% CI 2-sided [0.84 to 2.52]

16. Secondary Outcome: Number of Participants Who Had Cesarean Delivery
Time Frame: delivery
Population: Data was missing for 1 participant in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 329
Participants | 67 | 63
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.79 to 1.46]

17. Secondary Outcome: Number of Participants Who Reported Side Effects
Description: Number of participants who reported any side effect, nausea, urticaria, and/or an issue at the injection site
Time Frame: Any time during pregnancy from randomization to delivery, a timeframe up to 20 weeks
Population: Data was missing for 1 participant in the treatment group and 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 326 | 328
Participants
  Any | 223 | 220
  Injection site | 217 | 209
  Urticaria | 10 | 2
  Nausea | 7 | 10
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Any side effect; Test type: Superiority or Other; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.92 to 1.13]
Statistical Analysis 2: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Injection site; Test type: Superiority or Other; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.93 to 1.17]
Statistical Analysis 3: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Urticaria; Test type: Superiority or Other; Risk Ratio (RR) = 5.03, 95% CI 2-sided [1.11 to 22.78]
Statistical Analysis 4: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Nausea; Test type: Superiority or Other; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.27 to 1.83]

18. Secondary Outcome: Number of Participants Meeting the Composite Adverse Perinatal Outcome and Components
Description: comprised of fetal or infant death, respiratory distress syndrome, intraventricular hemorrhage (grades 3 and 4), periventricular leukomalacia, necrotizing enterocolitis (stage II and III), Bronchopulmonary dysplasia /chronic lung disease, retinopathy of prematurity (stage III or higher), early onset sepsis
Time Frame: within 72 hours of delivery
Population: With the exception of the composite outcome and death, the neonatal outcomes were only measured for live births.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Participants
  Composite Outcome Total | 23 | 30
  Fetal Death | 4 | 1
  Neonatal Death | 6 | 8
  Respiratory Distress Syndrome: number analyzed (Participants) | 320 | 323
  Respiratory Distress Syndrome | 13 | 16
  Bronchopulmonary dysplasia: number analyzed (Participants) | 320 | 322
  Bronchopulmonary dysplasia | 3 | 5
  Necrotizing enterocolitis, grade II or III: number analyzed (Participants) | 320 | 322
  Necrotizing enterocolitis, grade II or III | 2 | 5
  Intraventricular Hemorrhage, Grade III or IV: number analyzed (Participants) | 320 | 322
  Intraventricular Hemorrhage, Grade III or IV | 2 | 1
  Periventricular Leukomalacia | 4 | 1
  Early-onset Sepsis: number analyzed (Participants) | 320 | 322
  Early-onset Sepsis | 3 | 11
  Retinopathy of prematurity, grade II or IV: number analyzed (Participants) | 320 | 322
  Retinopathy of prematurity, grade II or IV | 1 | 3
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Analysis is for the total composite; Test type: Superiority or Other; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.46 to 1.30]

19. Secondary Outcome: Mean Birth Weight
Description: Birth weight as measured in grams
Time Frame: Delivery
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 327 | 330
Grams | 2855 (747) | 2824 (807)
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Birth Weight by Count of Participants
Description: Birth weight by count of participants < 2500 grams and < 1500 grams
Time Frame: Delivery
Population: Data was missing for 4 participants in the treatment group and 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 323 | 328
Participants
  Birth weight < 2500g | 72 | 75
  Birth weight < 1500g | 23 | 29

21. Secondary Outcome: Number of Neonates Who Measured Small for Gestational Age
Description: Birth weight percentile and small for gestational age <10th percentile based on number of weeks and gender.
Time Frame: Delivery
Population: Data was missing for 4 participants in the treatment group and 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 323 | 328
Participants
  < 10th percentile | 54 | 47
  < 3rd percentile | 15 | 14

22. Secondary Outcome: Number of Participants With Apgar Score of Less Than 7 at 5 Minutes
Description: The Apgar score is a simple method of quickly assessing the health and vital signs of a newborn baby created by and named after Dr. Virginia Apgar. Apgar testing assesses Appearance, Pulse, Grimace and Activity in a newborn and is typically done at one and five minutes after a baby is born, and it may be repeated at 10, 15, and 20 minutes if the score is low. The five criteria are each scored as 0, 1, or 2 (two being the best), and the total score is calculated by then adding the five values obtained. Agar scores of 0-3 are critically low, 4-6 are below normal, and indicate that the baby likely requires medical intervention, scores of 7+ are considered normal. The lower the Apgar score, the more alert the medical team should be to the possibility of the baby requiring intervention. Some components of the Apgar score are subjective, and there are cases in which a baby requires urgent medical treatment despite having a high Apgar score.
Time Frame: 5 minutes post delivery
Population: Data was missing for 4 participants in the treatment group and 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 323 | 328
Participants | 15 | 19

23. Secondary Outcome: Number of Neonates With a Major Congenital Anomaly
Description: Presence of a major congenital anomaly at birth
Time Frame: Delivery
Population: Data was missing for 1 participant in the treatment group and 2 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 326 | 328
Participants | 6 | 2

24. Secondary Outcome: Number of Neonates With Patent Ductus Arteriosus
Description: Number of neonates diagnosed with the heart defect patent ductus arteriosus
Time Frame: Delivery through neonatal discharge
Population: Data was missing for 7 participants in the treatment group and 8 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 320 | 322
Participants | 2 | 8

25. Secondary Outcome: Number of Neonates Experiencing Seizures
Description: Number of neonates experiencing seizures from delivery to hospital discharge
Time Frame: Delivery through neonatal discharge
Population: Data was missing for 7 participants in the treatment group and 8 participants in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 320 | 322
Participants | 1 | 2

26. Secondary Outcome: Number of Neonates Admitted to NICU
Description: Admission to the neonatal intensive care unit
Time Frame: Delivery through hospital discharge
Population: Data was missing for 5 participants in the treatment group and 1 participant in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 322 | 329
Participants | 63 | 69

27. Secondary Outcome: Median Length of NICU Stay
Description: Median length of stay in the neonatal intensive care unit in days
Time Frame: NICU admission through NICU discharge
Population: Data was missing for 5 participants in the treatment group and 1 participant in the placebo group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Number analyzed (Participants) | 322 | 329
days | 17 [6 to 43] | 15.5 [6 to 57.5]
Statistical Analysis 1: Comparison: 17 Alpha-hydroxyprogesterone Caproate vs Placebo; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the study period of April 2007 through June 2010, from the time of the participants randomization through hospital discharge of the mother and baby (up to 60 days).
Description: Other adverse events that are related to side effects are available for patients who had at least 1 study visit. 1 randomized participant in the treatment group and 2 randomized participants in the placebo group did not attend a study visit after randomization. Therefore the Ns for other side effects are different than those for the serious adverse events and the study sample (by 3 participants total).
Arm/Group | 17 Alpha-hydroxyprogesterone Caproate | Placebo
Serious Adverse Events (participants affected / at risk) | 22/327 | 13/330
Other Adverse Events (participants affected / at risk) | 326/326 | 328/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 17 Alpha-hydroxyprogesterone Caproate (N=327) | Placebo (N=330)
Miscarriage or stillbirth (Pregnancy, puerperium and perinatal conditions) | 5 | 1 — Miscarriage, antepartum stillbirth, intrapartum stillbirth
Placental abruption (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Pregnancy Complications (Pregnancy, puerperium and perinatal conditions) | 3 | 3 — advanced cervical dilation, oligohydramnios, preterm rupture of the membranes
Chest Pain (Vascular disorders) | 1 | 0
Epistaxis (Vascular disorders) | 1 | 0 — Nosebleed
Maternal Pulmonary edema (Cardiac disorders) | 1 | 0 — due to anemia and cardiac insufficiency
Maternal blood disorders (Blood and lymphatic system disorders) | 2 | 0 — Pulmonary embolism, thrombocytopenia
Congenital Anomalies (Congenital, familial and genetic disorders) | 5 | 3 — ovarian cyst, esophageal atresia, flexion contracture, hypospadias, patent ductus arteriosis, polydactyly, torticollis, Trisomy 21
Neonatal death (General disorders) | 6 | 8
Neonatal Hematochromatosis (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 17 Alpha-hydroxyprogesterone Caproate (N=326) | Placebo (N=328)
Headache (General disorders) | 7 | 8
Fatigue (General disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 7 | 10
Vomiting (Gastrointestinal disorders) | 6 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 6
Reaction at injection site (Skin and subcutaneous tissue disorders) | 217 | 210
Sore/burn at injection site (Skin and subcutaneous tissue disorders) | 145 | 153
Itching at injection site (Skin and subcutaneous tissue disorders) | 121 | 109
Swelling/lump at injection site (Skin and subcutaneous tissue disorders) | 107 | 93
Bruising at injection site (Skin and subcutaneous tissue disorders) | 26 | 23
Redness at injection site (Skin and subcutaneous tissue disorders) | 8 | 11
Urticaria (Skin and subcutaneous tissue disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No